CLINICAL TRIAL: NCT04159831
Title: A Phase 2, Randomized, Placebo-controlled, Double-blind, Dose-ranging Study Evaluating LTI-01 (Single-chain Urokinase Plasminogen Activator, scuPA) in Patients With Infected, Non-draining Pleural Effusions
Brief Title: A Study to Evaluate LTI-01 in Patients With Infected, Non-draining Pleural Effusions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rein Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LTI-01-2001
Record Dates: First submitted 2019-11-04; First posted 2019-11-12 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Pleural Effusion
MeSH Terms: conditions — Pleural Effusion | interventions — fibrinolytic agent LTI-01

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 400,000 U LTI-01 (Experimental): 400,000 U LTI-01 once a day (qd) x 3 days administered intrapleurally
  Interventions: Drug: LTI-01
- 800,000 U LTI-01 (Experimental): 800,000 U LTI-01 qd x 3 days administered intrapleurally
  Interventions: Drug: LTI-01
- 1,200,000 U LTI-01 (Experimental): 1,200,000 U LTI-01 qd x 3 days administered intrapleurally
  Interventions: Drug: LTI-01
- Placebo (Placebo Comparator): placebo (normal saline) 6ml qd x 3 days administered intrapleurally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LTI-01 — single-chain urokinase plasminogen activator, scuPA
  Arms: 1,200,000 U LTI-01; 400,000 U LTI-01; 800,000 U LTI-01
Drug: Placebo — normal saline
  Arms: Placebo

SUMMARY:
The LTI-01-2001 study is a double-blind, placebo-controlled, Phase 2 study to evaluate LTI-01 (single-chain urokinase plasminogen activator, scuPA) in patients with infected, non-draining pleural effusions.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female ≥ 18 years of age who provide written informed consent
* Clinical presentation compatible with complicated parapneumonic pleural effusion (CPE), empyema or other type of pleural infection
* Has pleural fluid requiring drainage as determined by chest ultrasonography or by chest CT, and which is either:
* a) purulent; b) gram stain positive; c) culture positive; d) pH < 7.2; or e) glucose < 60 mg/dL (3.3 mmol/L)
* Failure to adequately drain pleural fluid ≥ 3 hours post insertion of patent chest tube within the pleural space, as evidenced by one or more of the following criteria:
* > 2 cm depth of fluid by ultrasound or CT
* < 80% drainage from chest radiograph obtained prior to chest tube insertion.

Key Exclusion Criteria:

* Current pleural infection already treated with intrapleural fibrinolytic therapy
* Evidence of ipsilateral fibrothorax (e.g. CT scan with > 0.5 cm visceral pleural thickening)
* History of multiple thoracenteses or thoracic surgical procedures within 3 months of screening
* Previous pneumonectomy on the side of the pleural effusion
* Current bilateral pleural infections
* Known non-expandable lung prior to this pleural infection
* Known or high clinical suspicion of a malignant pleural effusion
* Existing indwelling or tunneled pleural catheter
* Current infected hepatic hydrothorax or evidence of another abdominal process (e.g. pancreatic cyst or renal cyst) communicating with the pleural space
* Active bleeding, or any condition in which bleeding is either a significant risk or would be difficult to manage
* Fully anticoagulated patients on heparin, warfarin or novel oral anti-coagulants who are not able to temporarily discontinue anti-coagulants while receiving study medication and for 2 days after last dose of study medication Note: patients receiving low-molecular weight heparin for immobilization or anti-platelet agents are not excluded.
* Presence of severe metabolic derangements that would interfere with study assessments
* Systolic blood pressure >185 mmHg or diastolic blood pressure > 110 mmHg at screening
* Hemodynamically unstable and/or requires use of intravenous vasopressor therapy
* Expected survival < 3 months from a pathology other than the qualifying infected, non-draining pleural effusion (e.g. metastatic lung carcinoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-09-26 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Incidence of referral to surgery | Post treatment (Day 4/Hospital discharge or at time of treatment failure)
  Treatment failure, as evidenced by continued or worsening pleural sepsis and failure to adequately drain pleural effusion, resulting in referral to surgery

SECONDARY OUTCOMES:
Relative change in pleural opacity | Post treatment (Day 4 or at time of treatment failure)
  Change from baseline in absolute pleural opacity and relative change from baseline in pleural opacity volume assessed by chest CT at Day 4

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - UC San Diego Health Jacobs Medical Center, La Jolla, California
  - University of California (UCLA), Los Angeles, California
  - UC Davis Medical Group, Sacramento, California
  - University of Colorado, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Rush University Medical Center, Chicago, Illinois
  - The University of Kansas Medical Center, Kansas City, Kansas
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. Luke's Health System, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - CHI CUMC Bergan Mercy, Omaha, Nebraska
  - North Shore - Long Island Jewish Medical Center, Queens, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - The Pennsylvania State University, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Vanderbilt Medical Center, Nashville, Tennessee
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas Health Science Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - INOVA, Fairfax, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No